CLINICAL TRIAL: NCT02599974
Title: Role of Fluorodeoxyglucose (FDG) PET-CT in the Initial Staging of Breast Cancer (ASAINT 1) and in the Early Assessment of Response to Neoadjuvant Chemotherapy (ASAINT 2)
Brief Title: PET-CT in the Initial Staging of Breast Cancer and in the Early Assessment of Response to Neoadjuvant Chemotherapy
Acronym: ASAINT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 12020 ASAINT
Record Dates: First submitted 2015-05-28; First posted 2015-11-09 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer; Positron-Emission Tomography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The two main objectives of this prospective study are:

* to identify those patients for whom pre-treatment FDG (Fluorodeoxyglucose) PET (positron emission tomography) CT-scan (Computed tomography scan) provides useful information for the treatment of breast cancer (ASAINT 1),
* to improve FDG PET-CT-scan imaging criteria for assessing response to neoadjuvant therapy early, in M0-patients (ASAINT 2).

The secondary objective is to better understand the interactions between the imaging parameters of FDG PET-CT-scan and biological and histological features of breast cancer .

This is a non-interventional study. Two PET-CT-scans are performed, one before starting treatment, and the other after 2 cycles of neoadjuvant chemotherapy. The two PET-CT-scans are prescribed by oncologists from the center of breast diseases Unit at St. Louis hospital, in Paris, France. Oncologists provide clear information to the patients on the purpose of the examination. The examinations are performed in the nuclear medicine department at St. Louis hospital. PET-CT-scans data, tumor characteristics, results of other imaging and biological tests, results of surgery and patient's follow-up are summarized in a "de-identified" file. This file has been declared to the National Commission on Informatics and Liberties (CNIL). The data in this file are established prospectively and secondary analyzed to assess the precise role of PET-CT-scans in the initial staging of breast cancer and to determine the optimal PET-CT-scans criteria to evaluate response to neoadjuvant treatment early.

ELIGIBILITY:
Inclusion Criteria :

* Histologically confirmed breast cancer
* Stage II and III breast cancer
* Neo-adjuvant chemotherapy
* Baseline PET-CT-scan (ASAINT 1 and 2)
* PET-CT-scans after second cycle of neo-adjuvant chemotherapy (ASAINT 2)
* Tumor biopsy for diagnosis and biological analysis with hormone receptors and Human Epidermal Growth Factor Receptor-2 (HER2) available
* Surgical intervention after completion of neo-adjuvant chemotherapy
* Evaluable pathological response

Exclusion Criteria :

* Other tumor localization
* Non controlled diabetes mellitus
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with large breast cancer treated with neo-adjuvant chemotherapy regimen.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2006-01; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response in M0 patients at baseline PET (stage II-III) | 18 weeks
  Absence of residual cancer cells in the primary breast tumor and in axillary lymph nodes

SECONDARY OUTCOMES:
Number of distant metastases (M1 patients at baseline PET) | 2 weeks
  Detection of distant metastases by FDG PET-CT
Number of metastatic nodes at baseline PET (axillary and extra-axillary) | 2 weeks
  Detection of metastatic axillary and extra-axillary nodes by FDG PET-CT
Standard uptake value on the FDG-PET (Fluorodeoxyglucose positron emission tomography) | 2 weeks
Patients overall survival | 5 years
event free survival | 5 years
Patients overall survival | 3 years
event free survival | 3 years
Patients overall survival | 2 years
event free survival | 2 years
Total lesion glycolysis on the FDG-PET (Fluorodeoxyglucose positron emission tomography) | 2 weeks
Metabolic tumor volume on the FDG-PET (Fluorodeoxyglucose positron emission tomography) | 2 weeks
Tumor heterogeneity determined on the FDG-PET (Fluorodeoxyglucose positron emission tomography) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Resche-Rigon, MD-PHD, Study Chair — DRCD APHP Paris; David Groheux, MD-PhD, Principal Investigator — APHP, IUH, University Paris Diderot, Paris 7, SPC
Locations (1):
- Hopital siant-Louis, Paris, Paris, France